CLINICAL TRIAL: NCT06460805
Title: axSEND: Exploring Immune and Microbiota Effects of a Partial Enteral Nutrition Diet in People With Axial Spondyloarthritis
Brief Title: axSEND: Exploring Immune and Microbiota Effects of a Partial Enteral Nutrition Diet in Axial Spondyloarthritis
Acronym: axSEND
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NHS Greater Glasgow and Clyde (Other)
Collaborators: University of Glasgow (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: GN23RH450
Record Dates: First submitted 2024-06-05; First posted 2024-06-14 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-06

CONDITIONS: Axial Spondyloarthritis; Ankylosing Spondylitis; Inflammation; Dysbiosis; Arthritis; Spondylitis; Spondylarthritis; SpA; AxSpA
Keywords: Partial Enteral Nutrition; Nutrition; Axial spondyloarthritis; Ankylosing spondylitis; axSpA; Diet; PEN; AS
MeSH Terms: conditions — Axial Spondyloarthritis; Spondylitis, Ankylosing; Inflammation; Dysbiosis; Arthritis; Spondylitis; Spondylarthritis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Axial Spondyloarthritis (Experimental)
  Interventions: Dietary Supplement: Partial enteral nutrition
- Healthy Volunteers (Experimental)
  Interventions: Dietary Supplement: Partial enteral nutrition

INTERVENTIONS:
Dietary Supplement: Partial enteral nutrition — 70% caloric intake from enteral nutrition formula and 30% caloric intake from a limited range of solid foods
  Other Names: PEN

SUMMARY:
People with axial spondyloarthritis (axSpA) often have intestinal inflammation and intestinal microbiome dysbiosis, with some similarities to Crohn's-like inflammatory bowel disease (IBD) gut inflammation. However, research has not addressed whether Partial Enteral Nutrition (PEN), a diet formed of a liquid formula and some solid whole foods, which is effective at inducing remission in IBD, may influence the dysbiotic microbiome and inflamed, hyperpermeable intestine of axSpA patients, and whether these changes may be accompanied by alterations in systemic markers of inflammation. Thus, there is a need to determine the effects of PEN on these aspects in axSpA patients.

In this study, the investigators intend to trial a 2-week course (with optional additional 2-week extension) of a PEN diet in people with active axSpA disease. A group of healthy volunteers following the same diet will act as a control.

ELIGIBILITY:
Eligibility Criteria for Participants with axSpA

Inclusion criteria. Participants will fulfil ALL of the following:

* Diagnosis of axSpA (fulfilling the ASAS criteria)
* Active disease (BASDAI score ≥4) on day of study visit
* Stable on treatment [defined as (1) no major change to therapy (change in treatment type) in the preceding 3 months AND (2) no minor change in therapy (adjustment of treatment dosage) in the preceding 1 month]
* Age ≥ 16 years
* Willing and able to give informed written consent.

Exclusion. Participants will have NONE of the following:

* Pregnancy or breastfeeding
* Prior diagnosis of IBD
* Recipient of chemotherapy/immunotherapy/radiotherapy in prior 3 months
* Recent systemic antibiotic use (within last 1 month)
* Current eating disorder
* Food allergy incompatible with diet (e.g. cow's milk allergy)
* Following a vegan diet
* Major surgery in prior 3 months or planned in forthcoming 3 months.
* Unable or unwilling to give informed consent
* Unable or unwilling to try the PEN diet.

Eligibility Criteria for Healthy Volunteer Participants

Inclusion criteria. Participants will fulfil ALL of the following:

* Age ≥ 16 years
* Current student and/or staff member at the University of Glasgow
* Willing and able to give informed written consent

Exclusion. Participants will have NONE of the following:

* Pregnancy or breastfeeding
* Prior diagnosis of an immune-mediated inflammatory condition
* Recipient of chemotherapy/immunotherapy/radiotherapy in prior 3 months
* Recent systemic antibiotic use (within last 1 month)
* Current eating disorder
* Food allergy incompatible with diet (e.g. cow's milk allergy)
* Following a vegan diet
* Major surgery in prior 3 months or planned in forthcoming 3 months.
* Unable or unwilling to give informed consent
* Unable or unwilling to try the PEN diet.

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2024-04-25 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Change in faecal butyrate at 2 weeks on a PEN diet | 2 weeks

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - NHS Greater Glasgow and Clyde, Glasgow
  - University of Glasgow, Glasgow

IPD SHARING:
Plan to Share IPD: No